CLINICAL TRIAL: NCT01184807
Title: A Phase 1, Open-label, Non-randomized, Dose-escalation Trial of OPB-51602 in Patients With Advanced Solid Tumors
Brief Title: Phase 1, Dose-escalation Trial of OPB-51602 in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Otsuka Beijing Research Institute (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 266-09-801-01
Record Dates: First submitted 2010-08-17; First posted 2010-08-19 (Estimated); Last update posted 2014-03-26 (Estimated); Status verified 2014-03

CONDITIONS: Malignant Solid Tumour
Keywords: Advanced solid tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- OPB-51602 (Other)
  Interventions: Drug: OPB-51602

INTERVENTIONS:
Drug: OPB-51602 — OPB-51602 at a dose of 2, 5, 10, 20, 40, 60, 80, or 100 mg/day,will be orally administered to subjects once daily for 2 weeks in each cycle of treatment in Dose Escalation Stage.A 2-day treatment-free interval will occur on Days 2 and 3 for PK sampling. Study drug administration will resume on Day 4 and continue until Day 17 in cycle 1.In Expansion stage part 1, OPB-51602 will be administered at recommend dose (4mg) for 3 weeks per cycle 9 2 weeks treatment and 1 week washout). There is also 2-day treatment free interval between Day 1 and Day 4 for PK sampling in cycle 1.In Expansion stage part 2, subject dosing will be started on Day 1 without 2-day treatment free interval and continued until Day 28 at recommend dose (4mg) first in Cycle 1. The same subjects will be treated at MTD(5mg)from cycle 2 onwards for 4 weeks per cycle.

SUMMARY:
This is an open-label, non-randomized, dose-escalation trial in patients with advanced solid tumors. The trial comprises 2 stages: a dose escalation stage at 8 dose levels of 2, 5, 10, 20, 40, 60, 80, and 100 mg/day,and possibly additional intermediate doses, to determine the MTD and recommended dose, and a subsequent 2 parts of expansion stage to investigate the safety profile and antitumor effect of OPB-51602 at the recommended dose.

DETAILED DESCRIPTION:
In expansion stage part 1, up to 20 advanced sold tumor subjects will be investigated the safety profiled and antitumor effect of OPB-51602 at the recommended dose for 3 weeks per cycle（2 weeks treatment and 1 week washout). In the expansion stage part 2, a maximum of 20 subjects with Non-small cell lung cancer (NSCLC), Melanoma or Gastrointestinal Stromal Tumor (GIST) will be treated until an investigational Medicinal product (IMP) efficacious case can be found. subject dosing will be started on Day 1 without 2-day treatment free interval and continued until Day 28 at recommend dose (4mg) first in cycle 1. After safety and tolerability are confirmed, same subjects will be treated at the MTD(5mg) from cycle 2 onwards as a once-daily oral dose for 4 weeks per cycle to obtain additional information about safety, tolerability and antitumor activity of OPB-51602

ELIGIBILITY:
Inclusion Criteria:

* Patients with pathologically confirmed, locally advanced or metastatic solid tumors who are unresponsive to standard therapy or for whom standard therapy is intolerable or unsuitable
* Age: ≥21 years (at time of informed consent)
* ECOG performance status: ≤2 (Appendix 1)
* Life expectancy of longer than 3 months
* Adequate vital organ function as follows:

  1. Bone marrow function Neutrophils: ≥1,500/μL, platelets: ≥75,000/μL, hemoglobin: ≥9.0 g/dL
  2. Hepatic function Aspartate transaminase (AST) and alanine transaminase(ALT): ≤2.5 ×institutional upper limit of normal(ULN) or ≤5.0 × institutional ULN if there is liver metastasis, serum total bilirubin: <2.5 × institutional ULN
  3. Renal function Serum creatinine: <1.5 × institutional ULN
* Capable of swallowing OPB-51602 tablets
* Ability to understand and willingness to sign written informed consent form (ICF) for participation in the trial
* No chemotherapy, radiotherapy, surgery, immunotherapy, or other therapy within 4 weeks prior to start of investigational medicinal product (IMP) administration and recovered from any prior toxicity
* If a subject has received more than 5 regimens of previous chemotherapy, the investigator must discuss with the sponsor regarding subject suitability prior to enrollment.

Exclusion Criteria:

* Uncontrolled central nervous system (CNS) metastasis
* Uncontrolled concurrent illness, including active infection, angina pectoris, cardiac arrhythmia, or heart failure (NYHA class III or IV, Appendix 2 New York Heart Association (NYHA) functional classification)
* Concurrent malignancy of a different type
* Immunocompromised subjects, including those who are known to be infected with human immunodeficiency virus (HIV)
* Psychiatric illness that would limit compliance with trial requirements
* Pregnant or breast-feeding women
* Women of childbearing potential (WOCBP) or male subjects whose partners are WOCBP who cannot or will not use effective contraceptive measures
* Administration of another investigational agent within 6 weeks prior to start of IMP administration
* Use of any of the prohibited medications and other substances listed in Appendix 3 CYP3A4 Inhibitors and Inducers within either 1 week prior to start of IMP administration or a period of at least 5 times the respective elimination halflife, whichever is longer
* Known severe gastrointestinal disorder, including malabsorption (at screening)
* Patients with CTCAE Grade 1 or higher pneumonitis (interstitial pneumonia) or pulmonary fibrosis* * If interstitial lung abnormalities, (e.g. ground-glass or linear opacity) are suspected on chest CT scan (high-resolution CT), regardless of whether or not there are any accompanying symptoms it must be confirmed, such as through consultation with a respiratory or radiology expert if necessary, that the patient dose not fall under this exclusion criterion before the patient can be enrolled in the trial.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2009-12; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
safety and tolerability | 3 weeks
  AEs, vital signs, body weight, ECG, clinical laboratory tests, and ECOG performances status in the first cycle of treatment

SECONDARY OUTCOMES:
Pharmacokinetics | duration of the treatment
  plasma and urinary concentrations of OPB-51602 and its metabolites
safety and tolerability | duration of treatment
  AEs, vital signs, body weight, ECG, clinical laboratory tests, and ECOG performances status in all treatment cycles.
efficacy | duration of treatment
  Response and progression evaluated using Response Evaluation criteria in solid tumors (RECIST)

CONTACTS AND LOCATIONS:
Overall Officials: Goh Boon Cher, Dr, Principal Investigator — Department of Haematology-Oncology,National University Hospital; Daniel Tan shao Weng, MD, PhD, Principal Investigator — National Cancer Centre, Singapore
Locations (2):
- Singapore (2):
  - National University Hospital (s) PTE LTD., Singapore, Singapore
  - National Cancer Centre, Department of Medical Oncology, Singapore

REFERENCES:
- [Derived] Wong AL, Soo RA, Tan DS, Lee SC, Lim JS, Marban PC, Kong LR, Lee YJ, Wang LZ, Thuya WL, Soong R, Yee MQ, Chin TM, Cordero MT, Asuncion BR, Pang B, Pervaiz S, Hirpara JL, Sinha A, Xu WW, Yuasa M, Tsunoda T, Motoyama M, Yamauchi T, Goh BC. Phase I and biomarker study of OPB-51602, a novel signal transducer and activator of transcription (STAT) 3 inhibitor, in patients with refractory solid malignancies. Ann Oncol. 2015 May;26(5):998-1005. doi: 10.1093/annonc/mdv026. Epub 2015 Jan 21. PMID 25609248